CLINICAL TRIAL: NCT06878625
Title: A Multicenter, Prospective, Cohort Study Evaluating the Efficacy of Trop-2 ADC Combination Therapy in Advanced Triple-Negative Breast Cancer
Brief Title: A Multicenter, Prospective, Cohort Study of Trop-2 ADC Combination Therapy for Advanced Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Chunfang Hao, Associate Chief Physician, Department of Breast Oncology, Tianjin Medical University Cancer Institute and Hospital, Tianjin Medical University Cancer Institute and Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y-Gilead2024-PT-0235
Record Dates: First submitted 2025-01-31; First posted 2025-03-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Evaluating the Efficacy of Trop-2 ADC Combination Therapy in Advanced Triple-Negative Breast Cancer
Keywords: Sacituzumab govitecan; triple negative breast cancer; PD-1 monoclonal antibody; anti-angiogenesis
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacituzumab govitecan combined with Toripalimab (Experimental): Sacituzumab govitecan (Trop-2 ADC) : 10mg/kg on days 1 and 8, intravenous infusion, every 3 weeks for a treatment cycle.
  Toripalimab 240 mg was given intravenously on day 1 of each cycle, every 3 weeks for a treatment cycle.
  Interventions: Combination Product: Sacituzumab Govitecan combined with Toripalimab
- Sacituzumab govitecan combined with anti-angiogenesis (Experimental): Sacituzumab govitecan (Trop-2 ADC) : 10mg/kg on days 1 and 8, intravenous infusion, every 3 weeks for a treatment cycle.
  Antiangiogenesis targeted drugs: Bevacizumab or Anlotinib Hydrochloride, according to the standard dose treatment.
  Interventions: Combination Product: Sacituzumab govitecan combined with anti-angiogenesis

INTERVENTIONS:
Combination Product: Sacituzumab Govitecan combined with Toripalimab — Sacituzumab Govitecan combined with Toripalimab
  Arms: Sacituzumab govitecan combined with Toripalimab
Combination Product: Sacituzumab govitecan combined with anti-angiogenesis — Sacituzumab govitecan combined with anti-angiogenesis( Bevacizumab or Anlotinib Hydrochloride)
  Arms: Sacituzumab govitecan combined with anti-angiogenesis

SUMMARY:
Research purposes: the research design in the late more than 2 lines TNBC prospective, multicenter, cohort study, respectively to observe Trop2 - ADC joint PD - 1 single or combined anti-angiogenesis drugs (macromolecular single bevacizumab or small molecules TKI resistance, for, as the default layered) the efficacy and safety. Indications: Trop2 - ADC joint PD - 1 single or combined anti-angiogenesis drugs (macromolecular single bevacizumab or small molecules TKI resistance, for, as the default layered) treat above 2 late three negative breast cancer (TNBC).

DETAILED DESCRIPTION:
1. Study Population

   - Eligible Participants: Patients with triple - negative metastatic breast cancer at the second line of treatment or higher. Triple - negative invasive breast cancer is histologically confirmed, defined as immunohistochemical detection revealing estrogen receptor (ER) < 10%, progesterone receptor (PR) < 10%, and HER2 0 - 1+ or HER2 2+ with negative fluorescence in situ hybridization (FISH) or chromogenic in situ hybridization (CISH) results, in accordance with the 2018 ASCO - CAP HER2 - negative identification guidelines.
2. Experimental Design

   - Study Type: Multicenter, prospective cohort study.
3. Sample Size Determination

   * The sample size is calculated based on the primary endpoint of progression - free survival (PFS). Drawing on data from ASCENT (a confirmatory phase III study on the efficacy in triple - negative breast cancer) and EVER - 132 - 001 (a Chinese population bridging study presented at the ESMO Congress), the PFS of sacituzumab govitecan monotherapy in metastatic triple - negative breast cancer (mTNBC) is approximately 5.6 months.
   * Assuming a hazard ratio of 0.70 in each cohort (median PFS value of 8 months vs. 5.6 months), to detect a statistically significant difference between the trial group and the sacituzumab govitecan monotherapy control group at a one - sided significance level of 0.05 and a power of 80%, 51 PFS events are required.

   Given an enrollment period of 18 months and a total study duration of 30 months, 69 subjects are needed for each cohort.
4. Dosage Regimens

   * 4.1 Sacituzumab Govitecan Dose and Administration: The recommended dose is 10 mg/kg. It is administered by intravenous infusion on days 1 and 8 of each treatment cycle, with each cycle lasting three weeks.
   * 4.2 Toripalimab Dose and Administration: 240 mg is administered by intravenous infusion on day 1 of each cycle. Each treatment cycle has a duration of three weeks.
   * 4.3 Antiangiogenic Targeted Drugs Options and Dosage: Bevacizumab or Anlotinib can be selected. Treatment is carried out according to the standard dosage for each respective drug.
5. Inclusion Criteria

   * Age between 18 and 70 years.
   * Histologically - confirmed triple - negative invasive breast cancer as per the defined immunohistochemical and molecular criteria.
   * For patients with locally advanced or metastatic breast cancer:

   Those who have undergone radical surgery. Those who have received at least one but no more than two lines of chemotherapy in the advanced treatment phase. Additionally, early - stage triple - negative breast cancer patients who experienced disease progression within one year after neoadjuvant or adjuvant therapy are eligible.
   * No prior use of immunotherapeutic drugs or anti - angiogenic drugs.
   * At least one measurable lesion as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
   * No contraindications to chemotherapy, immunotherapy, or anti - angiogenic therapy.
   * Permitted to have stable or asymptomatic brain metastases.
   * Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 - 2, with a predicted survival exceeding 12 weeks.
   * All acute toxicities from previous anticancer therapies must have resolved to Grade ≤1 according to the protocol criteria (excluding alopecia) before screening.
   * Women of childbearing potential must agree to use medically approved contraception during treatment and for at least three months post - treatment.
   * Adequate organ function meeting the following criteria:

   Hemoglobin ≥ 90 g/L without transfusion within 14 days. Absolute Neutrophil Count (ANC) ≥ 1.5×10⁹/L. Platelets ≥ 75×10⁹/L. Total Bilirubin ≤ 1.5× the upper limit of normal (ULN). Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3×ULN (≤ 5×ULN if liver metastasis is present).

   Serum Creatinine ≤ 1×ULN. Left Ventricular Ejection Fraction (LVEF) ≥ 50%.

   - Participants must voluntarily enroll in the study, demonstrate excellent adherence, and actively participate in safety and survival follow - up assessments.
6. Exclusion Criteria

   * Uncontrolled central nervous system metastases (symptomatic or requiring glucocorticoids or mannitol for symptom management).
   * Symptomatic third - space effusions, including pericardial, pleural, and peritoneal effusions, that cannot be adequately managed by drainage or other therapeutic interventions.
   * Participation in another clinical trial within 30 days prior to enrollment. History of other malignancies within the past 5 years, excluding adequately treated cervical carcinoma in situ, skin squamous cell carcinoma, thyroid carcinoma, or controlled basal cell carcinoma.
   * Uncontrolled cardiac conditions, including:
   * Heart failure classified as NYHA class II or higher.
   * Unstable angina.
   * Myocardial infarction within the past year.
   * Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
   * QTc interval greater than 470 ms.
   * Arterial or venous thrombotic events within 24 weeks preceding informed consent, such as cerebrovascular accidents (e.g., transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
   * Within 24 weeks prior to signing the informed consent form (ICF), a history of any of the following conditions: peptic ulcer, gastrointestinal perforation, corrosive esophagitis or gastritis, inflammatory bowel disease, diverticulitis, abdominal fistula, tracheoesophageal fistula, or intra - abdominal abscess.

   Presence of factors that significantly impair oral drug absorption, such as inability to swallow, chronic diarrhea, or intestinal obstruction.
   * Documented history of allergy with potential hypersensitivity or intolerance to sacituzumab govitecan, toripalimab, bevacizumab, or anlotinib.
   * Active human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B surface antigen positive and HBV DNA ≥ 500 IU/ml), or hepatitis C (hepatitis C antibody positive and detectable HCV RNA).
   * Pregnant women, lactating women, fertile women with a positive baseline pregnancy test, or women of childbearing age who are unwilling to use effective contraception for the duration of the trial.
   * Presence of concomitant diseases (e.g., poorly controlled hypertension, severe diabetes, neurological or psychiatric disorders) or any other condition that, in the investigator's judgment, could compromise subject safety, confound study results, or prevent subjects from completing the study.
7. Efficacy Endpoints

   * 7.1 Primary Endpoint Progression - free survival (PFS).
   * 7.2 Secondary Endpoints Objective response rate (ORR). Overall survival (OS). Safety evaluation. Duration of response (DOR). Clinical benefit rate (DCR). Biomarker studies.
   * Efficacy is evaluated every two cycles. For treatments showing effectiveness (at least 4 to 6 cycles), immunotherapy or targeted therapy can be continued.
8. Safety Indicators

   - Adverse events are recorded from the time of completion or signing of the informed consent until the end of the study period as determined by the researchers. All adverse events occurring during this period are to be documented.
9. Statistical Methods

   * 9.1 General Data Summarization：Unless otherwise specified, data will be summarized using descriptive statistical methods. For measurement data, the mean, standard deviation, median, maximum, and minimum values will be reported. For count data, frequencies and percentages will be used for summarization.
   * 9.2 Survival Analysis：The Kaplan - Meier method will be employed to estimate survival rates and plot survival curves for time - to - event data, such as PFS and DOR.
   * 9.3 Blood Concentration Data：Blood concentration data will be summarized using the geometric mean, geometric standard deviation, geometric coefficient of variation, mean, standard deviation, coefficient of variation, median, maximum, and minimum values.
   * 9.4 Effectiveness Analysis： Effectiveness analysis will be based on the full analysis set (FAS) and the per - protocol set (PPS).The objective response rate (ORR) will be descriptively statistically analyzed according to the stage and dose groups. The number and proportion of subjects with a response (complete response (CR)+partial response (PR)) will be provided, and a two - sided 95% exact confidence interval for the overall ORR will be estimated.PFS and DOR, being time - to - event data, will be analyzed using the Kaplan - Meier method to plot survival curves and estimate the median survival time. When necessary, the two - sided 95% confidence interval for the overall median survival time will be estimated.The clinical benefit rate (DCR) will provide the number and proportion of subjects identified as CR + PR+stable disease (SD), and when necessary, a two - sided 95% exact confidence interval for the DCR will be estimated.
   * 9.5 Safety Analysis：Safety analysis will be based on the safety set (actual drug categories). It is limited to summary descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years.
2. Histologically confirmed triple-negative invasive breast cancer, defined as immunohistochemical detection of ER < 10%, PR < 10%, HER2 0-1+ or HER2 2+ with negative FISH or CISH results, in accordance with the 2018 ASCO-CAP HER2-negative identification guidelines.
3. Patients with locally advanced or metastatic breast cancer who have undergone radical surgery; patients received at least one but no more than two lines of chemotherapy in the advanced treatment phase. Early-stage triple-negative breast cancer patients who experienced disease progression within one year after neoadjuvant or adjuvant therapy are also eligible.
4. No prior use of immunotherapy or anti-angiogenic drugs.
5. At least one measurable lesion based on RECIST 1.1 criteria.
6. No contraindications to chemotherapy, immunotherapy, or anti-angiogenic therapy.
7. Stable or asymptomatic brain metastases are permitted.
8. ECOG Performance Status (PS) score of 0-2; predicted survival exceeding 12 weeks.
9. All acute toxicities from previous anticancer therapies must have resolved to Grade ≤1 per protocol criteria (excluding alopecia) before screening.
10. Women of childbearing potential must agree to use medically approved contraception during treatment and for at least three months post-treatment.
11. Adequate organ function, meeting the following criteria: Hemoglobin ≥90 g/L without transfusion within 14 days; Absolute Neutrophil Count (ANC) ≥1.5×10^9/L; Platelets ≥75×10^9/L; Total Bilirubin ≤1.5×ULN; AST and ALT ≤3×ULN (≤5×ULN if liver metastasis present); Serum Creatinine ≤1×ULN; Left Ventricular Ejection Fraction (LVEF) ≥50%.
12. Participants were voluntarily enrolled in this study, demonstrated excellent adherence, and actively participated in safety and survival follow-up assessments.

Exclusion Criteria:

1. Uncontrolled central nervous system metastasis (symptomatic or requiring glucocorticoids or mannitol for symptom management);
2. Symptomatic third-space effusions, including pericardial, pleural, and peritoneal effusions, that cannot be adequately managed by drainage or other therapeutic interventions;
3. Participation in another clinical trial within 30 days prior to enrollment;
4. History of other malignancies within the past 5 years, excluding adequately treated cervical carcinoma in situ, skin squamous cell carcinoma, thyroid carcinoma, or controlled basal cell carcinoma;
5. Uncontrolled cardiac conditions, such as: (1) heart failure classified as NYHA class II or higher; (2) unstable angina; (3) myocardial infarction within the past year; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; (5) QTc interval greater than 470 ms;
6. Arterial or venous thrombotic events within 24 weeks preceding informed consent, including cerebrovascular accidents (e.g., transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
7. Within 24 weeks prior to signing the informed consent form (ICF), a history of any of the following conditions: peptic ulcer, gastrointestinal perforation, corrosive esophagitis or gastritis, inflammatory bowel disease, diverticulitis, abdominal fistula, tracheoesophageal fistula, or intra-abdominal abscess.
8. Presence of factors that significantly impair oral drug absorption, such as inability to swallow, chronic diarrhea, or intestinal obstruction.
9. Patients with a documented history of allergy may have potential hypersensitivity or intolerance to gozzatuzumab, toripalimab, bevacizumab, or anlotinib.
10. Active infection with human immunodeficiency virus (HIV), active hepatitis B (hepatitis B surface antigen positive and HBV DNA ≥500 IU/ml), or hepatitis C (hepatitis C antibody positive and detectable HCV RNA).
11. Pregnant women, lactating women, fertile women with a positive baseline pregnancy test, or women of childbearing age who are unwilling to use effective contraception for the duration of the trial.
12. Presence of concomitant diseases (e.g., poorly controlled hypertension, severe diabetes, neurological or psychiatric disorders) or any other condition that, in the investigator's judgment, could compromise subject safety, confound study results, or prevent subjects from completing the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Until progression or death, up to approximately 60 months
  PFS is defined as time from date of randomization until the date of first objective progressive disease (PD) by investigator assessment according to RECIST v1.1 or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Investigator per RECIST Version 1.1 | Until progression, up to approximately 60 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.
Overall Survival (OS) | Until death, up to approximately 60 months
  OS is defined as the time from randomization until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided